CLINICAL TRIAL: NCT05808153
Title: Innovative Imaging and Cognitive BIOmarkers to Predict Huntington's Disease Progression
Acronym: I2BIO-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP210360; 2021-004141-20 (EudraCT Number)
Record Dates: First submitted 2022-12-15; First posted 2023-04-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-01

CONDITIONS: Huntington Disease
Keywords: Huntington's disease; Biomarkers; Cognition; Disease progression; Imaging
MeSH Terms: conditions — Huntington Disease; Disease Progression

STUDY DESIGN:
Intervention Model Description: Model description: Identification, evaluation and validation of new clinical, biological and imaging biomarkers (MRI without contrast product and PET with intravenous administration of a radiotracer) on a prospective cohort of carriers of the mutation responsible for Huntington's disease and healthy volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic (MH) and pre-symptomatic (preMH) patients (Experimental): * Number of GAC ≥ 40
  * GAP score ≥ 250
  * 10 ≤ TFC ≤ 13
  * TMS >5 if TFC=13
  * Diagnostic confidence level =4
  * Age onset of the disease > 20 years
  * Patients in physical capacity to sign the consent
  Interventions: Radiation: radiotracer injection
- Age-matched controls (healthy volunteers) (Active Comparator): * TFC functional UHDRS score = 13
  * TMS engine UHDRS rating < 6
  Interventions: Radiation: radiotracer injection

INTERVENTIONS:
Radiation: radiotracer injection — MRI with radiotracer injection

SUMMARY:
Intro Huntington's disease (HD) patients suffer from motor, cognitive and behavioral impairments, with heterogeneous phenotypes and variable time course. This leads to a high variance of HD markers, none of which is currently sensitive enough to 1) measure disease progression from small cohort data, 2) predict disease entry in carriers of the HD mutation (during the prodromal phase or in patients considered asymptomatic: pre-HD patients), and 3) measure a significant evolution of the state of pre-HD patients over a time window compatible with the realization of clinical trials (about 2/3 years). Moreover, the markers of HD do not allow a fine stratification of the patients.

Hypothesis/Objective Our objectives are 1) to evaluate the sensitivity of new markers and assessment tools for symptomatic (HD) and presymptomatic (pre-HD) patients, 2) to define a model of disease progression, and 3) to establish an enrichment strategy to improve patient selection for future therapeutic trials.

Method We will evaluate newly developed cognitive tests, multimodal imaging techniques, biological markers and use innovative statistical approaches.

We will follow 60 patients with the mutation responsible for MH (40 presymptomatic pre-MH patients, 20 symptomatic MH patients) and 20 healthy volunteers (controls) over a 24-month period.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:
* Age ≥18 years and ≤65 years
* Information and collection of written consent
* Affiliation with a social security plan, beneficiary or beneficiary's right
* Healthy controls
* UHDRS functional score TFC = 13
* Motor UHDRS score TMS < 6 With no known genetic disease and no direct relationship to an HD patient or family ancestors carrying the HD mutation (or knowing their genetic status with CAG < 36).
* Manifest carriers
* Number of GACs ≥ 40
* CAP score ≥ 250
* 10 ≤ TFC ≤ 13
* TMS >5 if TFC=13
* Diagnostic confidence level =4
* Age of onset of disease > 20 years
* Patients physically able to sign consent
* Premanifest carriers
* Number of GACs ≥ 40
* CAP score ≥250
* CFT = 13
* TMS < 6
* Patients physically able to sign consent

Exclusion Criteria:

* Participant under guardianship or curatorship
* Neurological or psychiatric disorder unrelated to HD
* Intercurrent illness that may impact participant's performance
* Chronic progressive neurological disease
* Claustrophobia
* Brain injury unrelated to HD
* Pacemaker, intracorporeal metal, intracerebral clip, any metallic foreign body: implantable cardiac electronic device such as pacemakers, implantable cardioverter defibrillators etc., metallic intraocular foreign bodies, implantable neurostimulation systems, cochlear implants/ear implants, drug infusion pumps (insulin administration, analgesic drugs), or chemotherapy pumps): if possible, the patient should remove the device.
* Catheters with metal components (Swan-Ganz catheter), metal fragments such as bullets, shotgun pellets and metal shrapnel, cerebral artery aneurysm clips, magnetic dental implants, tissue expander, artificial limb, hearing aid, piercing such as pacemaker,
* Known hypersensitivity to the radiopharmaceutical preparation (excipients in the radiopharmaceutical preparation)
* Pregnant or breastfeeding woman
* Person under state medical aid
* Person deprived of liberty
* Person participating or having participated in an interventional study for less than 3 months or without time limit in a trial of neural transplants or gene therapy.
* Person participating or having participated in a research protocol with a radiopharmaceutical injection for less than 12 months.
* Neurological or psychiatric disorder unrelated to HD
* Intercurrent disease that may impact participant's performance
* Chronic progressive neurological disease
* Claustrophobia
* Brain injury unrelated to HD
* Pacemaker, intracorporeal metal, intracerebral clip
* Pregnant, breastfeeding or wanting to procreate during participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-04-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Genetic markers | Visit Month 0

SECONDARY OUTCOMES:
cognitive tests | Visits Month 0, Month 1, Month 12, Month 24
  Cognitive scores - Neurological scores- Psychiatric scores
biological markers | Visits Month 0, Month 1, Month 12, Month 24
  Neuroinflammation markers in blood - Neurodegeneration markers in blood
multimodal imaging techniques | Visits Month 0, Month 12, Month 24
  MRI
multimodal imaging techniques | Visits Month 0, Month 24
  PET/MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Henri MONDOR, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided